CLINICAL TRIAL: NCT06727019
Title: Daily Low-level Red Light and 0.01% Low-dose Atropine for Myopia Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, cao kai, Dr, Beijing Tongren Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BeijingTH2023qiao
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- red-light (Experimental): In the low-level red-light (LLRL) group, the children used LLRL irradiation twice a day for 3-minute sessions, ensuring a gap of over 4 h between each use
  Interventions: Device: low-level red-light
- atropine (Experimental): participants in the atropine group used 0.01% low-dose atropine eye drops once each night
  Interventions: Drug: Atropine (0.01%)

INTERVENTIONS:
Device: low-level red-light — 650-nm low-level red-light
  Arms: red-light
Drug: Atropine (0.01%) — Atropine eye drops at concentration of 0.01%
  Arms: atropine

SUMMARY:
To compare the preventive effects of daily low-level red-light and 0.01% low-dose atropine eye drops on myopia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged at least 7 years old. 2. The spherical equivalent error (SER) after pupil dilation was between -0.5 D and +0.75D.

  3. Had a record of cycloplegia SER at least 6 months before this study, and SER changed -0.5D compared with the last measurement or had a family history of high myopia.

  4. Corneal astigmatism ≤ 1.25D. 5. Interocular refraction discrepancy ≤ 1.5D. 6. No allergy history of cycloplegia drugs. 7. Willingness to participate in the study and signed informed consent.

Exclusion Criteria:

- 1. Intraocular pressure was below 10 mm Hg or higher than 22 mm Hg. 2. Presence of amblyopia, or ocular pathological conditions such as retinal, lens, or corneal disorders.

3. Children currently using other myopia interventions other than LDA or LLRL. 4. Children with systemic and immune disorders, such as albinism, psoriasis, nephrotic syndrome, systemic lupus erythematosus, and diabetes 5. Individuals with conditions like Tourette's syndrome or epilepsy.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of myopia | 12 months
  12-month incidence of myopia

CONTACTS AND LOCATIONS:
Overall Officials: Liya Qiao, PhD, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data would be avialable on reasonable request